CLINICAL TRIAL: NCT04002102
Title: Open-Label Placebos to Treat Fatigue in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tapan Shirish Mehta, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300003575
Record Dates: First submitted 2019-06-25; First posted 2019-06-28 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: Placebo; Open-Label
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — Glucose; Standard of Care; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OLP treatment (Experimental): Participants randomized to the treatment group will receive: 1) educational materials; 2) positive expectancy; 3) 2 placebo pills twice a day for 21 days.
  Interventions: Other: OLP treatment
- Usual care (Other): Participants randomized to the no treatment group will remain in standard care alone for 21 days and receive educational materials.
  Interventions: Other: Usual care
- Expectancy Group (Active Comparator): Participants receive educational materials and positive expectancy orientation via Zoom or telephone
  Interventions: Other: Expectancy Group

INTERVENTIONS:
Other: OLP treatment — Receive two open-label placebo pills twice a day after randomization. Will receive for 21 days and then stop. It will include educational materials and positive expectancy.
  Other Names: Open-Label placebo; Glucose Tablet
  Arms: OLP treatment
Other: Usual care — Remain in standard care after randomization and educational materials.
  Other Names: Standard care
  Arms: Usual care
Other: Expectancy Group — Educational materials and positive expectancy orientation via Zoom or telephone
  Other Names: Education
  Arms: Expectancy Group

SUMMARY:
Fatigue is one of the most prevalent and disabling symptoms of multiple sclerosis. Current treatments, including pharmacological, physical therapy, sleep regulation and psychological interventions are of marginal benefit. Pharmacological treatments have inconsistent evidence. Recent studies show that non-deceptive open-label placebos (OLP) have moderate-to-large effects on symptoms, including fatigue, in adults with a variety of medical conditions.

Hence, this is a pilot and feasibility study to obtain data on the feasibility and effects of OLP for multiple sclerosis related fatigue and its impact to provide the basis for a competitive NIH application. This pilot study will be the first study to evaluate whether OLP, that garners full consent and engages patients in their wellness, may offer a safe, effective treatment for multiple sclerosis related fatigue.

DETAILED DESCRIPTION:
The purpose of this pilot study is to evaluate the feasibility of recruiting, enrolling and retaining participants in a study on the acceptability and effects of a non-deceptive (open-label) administration of placebo pills for treating MS related fatigue. Specific Aim 1 will assess the feasibility endpoints including accrual (enroll 44 participants), retention (80% of the sample) and placebo adherence (90%). Specific Aim 2 will evaluate the between-group changes in fatigue, quality of life, cognitive functioning and self-efficacy. Specific Aim 3 will evaluate participant acceptability, satisfaction and experience.

Design:

This pilot study is a randomized control trial consisting of three arms: open label placebo arm, expectancy arm, and usual care arm. The clinical coordinator will review medical records, enroll and consent participants based on the following inclusion criteria: diagnosis of MS, 19 years or older, report of moderate to severe fatigue, PDDS score of < 7, and stable dose of DMTs for 90 days.

Exclusion criteria consists of: major comorbid conditions and use of off label medications or exercise programs in the past 30 days, and if one is confined to a wheelchair.

Baseline and 21 day tele assessments will involve objective measures performed by a physical therapist, Single Digit Modality Test (SDMT) and Five Time Sit to Stand (FTSST) and subjective questionnaires sent to participant's email including Modified Fatigue Impact Scale (MFIS), Functional Systems Score (FSS), Patient Reported Outcomes Measurement Information System (PROMIS), Perceived Deficits Questionnaire, Epworth Sleepiness Scale, and the SF-36 assess of quality of life. Participants will be randomized by the clinical coordinator after baseline testing. The open label placebo and expectancy arm will meet with the care provider who will follow a scripted orientation that mimics a typical patient-provider interaction when prescribing a medication, including the rationale for effectiveness. The provider will emphasize the importance of adherence to the medication for the open label placebo arm and the breathing exercises for the expectancy arm for the next 21 days. A tracking sheet will be provided to both arms to document adherence. The usual care arm will meet with the care provider who will follow a scripted orientation on fatigue and heat management strategies. All participants will receive educational materials on fatigue and heat management. A day 11 check in call will be made to gauge progress and answer questions. After the 21 day tele assessment is performed, the participant will complete subjective questionnaires via email for 28 day and 35 day follow up.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of MS
* Aged 19 years or older
* report moderate-to-severe fatigue (i.e., ≥4 on the FSS)
* Patient Determined Disease Steps score of ≥7.

Exclusion Criteria:

* Major comorbid conditions that might influence fatigue (e.g. lupus, chronic fatigue syndrome)
* Patients treated with off label medications or exercise program in the past 30 days.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline fatigue at 21 days using the Fatigue Severity Scale (FSS). | Participants will complete this scale at baseline and 21 days later, the participant will spend 10 minutes each assessment completing this scale.
  This scale is used to measure fatigue and the scale has a range from 9-63 with 9 being the best possible score and 63 being the worst score.
Change from baseline impact of fatigue at 21 days using the Modified Fatigue Impact Scale (MFIS). | Participants will complete this scale at baseline and 21 days later, the participant will spend 15 minutes each assessment completing this scale.
  This scale is used to measure fatigue and the scale has a range from 0 to 84 with 0 being the best possible score and 84 being the worst score.
Change from baseline quality of life at 21 days using the 36-item Short Form survey (SF-36). | Participants will complete this scale at baseline and 21 days later, the participant will spend 15 minutes each assessment completing this scale.
  The scores for this survey range from 0-100 with 0 being the worst possible score and 100 being the best possible score.

SECONDARY OUTCOMES:
Change from baseline sleepiness at 21 days using the Epworth Sleepiness Scale (ESS). | Participants will complete this scale at baseline and 21 days later, the participant will spend 15 minutes each assessment completing this scale.
  This scale is used to measure sleepiness and the scale has a range from 0-24 with 0 being the best possible score and 24 being the worst.
Change from baseline neurological functioning at 21 days using the Perceived Deficit Questionnaire 5-Item Version (PDQ-5). | Participants will complete this scale at baseline and 21 days later, the participant will spend 15 minutes each assessment completing this scale.
  The scores for this questionnaire range from 5-25 with 5 being the best possible score and 25 being the worst possible score.
Godin Leisure-Time Exercise Questionnaire | Participants will complete this scale at baseline and 21 days later
  A self-explanatory, brief four-item query of usual leisure-time exercise habits

OTHER OUTCOMES:
Change from baseline general self efficacy for managing chronic conditions at 21 days using the PROMIS instrument | Participants will complete this scale at baseline and 21 days later, the participant will spend 15 minutes each assessment completing this scale.
  The scores for this tool are coded separately for each of the 10 questions and range from 1-5 for questions Global01-06, 08r, 09r, and 10r with 1 being the worst possible score and 5 being the best possible score and a range from 0-10 for question Global07r with 0 being the worst possible score and 10 being the best possible score.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan S Mehta, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Tanner Foundation, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: Yes
To be determined. Sharing study protocol, statistical analysis plan, and informed consent.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will be posted on CT.gov
Access Criteria: To be determined

REFERENCES:
- [Derived] Baidwan NK, Tracy T, Chiu CY, Nawshin T, Hoenemeyer T, Riser E, Motl R, Fontaine K, Mehta T. Open label placebo to treat fatigue in people with multiple sclerosis: feasibility and preliminary effects. Pilot Feasibility Stud. 2025 Jul 3;11(1):93. doi: 10.1186/s40814-025-01674-w. PMID 40611184